CLINICAL TRIAL: NCT00960505
Title: Alternate Day Fasting for Weight Loss, Weight Maintenance and Cardio-protection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Pennington Biomedical Research Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Krista Varady, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-0118; R01HL106228 (NIH)
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Coronary Heart Disease; Obesity; Weight Loss
Keywords: Diet; Coronary heart disease; Obesity; Weight loss; Weight maintenance
MeSH Terms: conditions — Coronary Disease; Obesity; Weight Loss | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alternate day fasting (ADF) (Experimental): Fast day diet: 25% energy intake, Feast day diet: Ad libitum energy intake (alternating days)
  Interventions: Other: Alternate day fasting
- Calorie restriction (CR) (Experimental): 75% energy intake every day
  Interventions: Other: Calorie restriction
- Control (Active Comparator): Usual diet
  Interventions: Other: Control diet

INTERVENTIONS:
Other: Alternate day fasting
  Arms: Alternate day fasting (ADF)
Other: Calorie restriction
  Arms: Calorie restriction (CR)
Other: Control diet
  Arms: Control

SUMMARY:
The proposed research will demonstrate that alternate day modified fasting (ADMF) is a suitable alternative to daily calorie restriction (CR) for weight loss, weight maintenance, and heart disease prevention. Since many overweight and obese individuals find it difficult to adhere to daily CR, this diet option may improve adherence with these dietary restriction protocols. This, in turn, will allow a greater percent of the overweight and obese population to lose weight, maintain weight loss, and prevent future occurrences of coronary heart disease.

DETAILED DESCRIPTION:
Overweight and obese individuals are at increased risk for coronary heart disease (CHD). Losing weight by means of dietary restriction greatly reduces vascular disease risk. The majority of studies examiningmost common dietary restriction protocol s implemented is daily calorie restriction (CR). Another dietary restriction regimen employed, although far less commonly, is alternate day modified fasting (ADMF). ADMF involves a "feed day" where food is consumed ad-libitum, alternated with a "fast day", where food intake is partially reduced. Previous reports show that adherence to ADMF exceeds that of CR after 8 weeks of treatment. This increased adherence to ADMF results in greater weight loss, which produces more pronounced improvements in CHD risk. What has yet to be determined is whether adherence to ADMF remains near maximal for longer treatment durations (24 weeks), and if this improved adherence results in greater reductions in body weight and CHD risk, versus CR. Once weight loss is achieved, weight maintenance is extremely important as CHD risk can increase if weight is regained. Whether ADMF is an effective strategy for weight maintenance remains unknown. Accordingly, the aims of this proposal are: Aim 1: To establish that adherence to ADMF is greater than that of CR during a 24-week intervention period and to determine if increased adherence to ADMF results in greater weight loss; Aim 2: To establish that greater reductions in body weight by ADMF over a 24-week period will result in greater improvements in traditional CHD risk parameters (blood pressure, plasma lipid levels, cholesterol synthesis rate, LDL particle size, and CRP) and emerging CHD risk parameters (fat cell-derived hormones, body fat distribution, and fat cell size) in comparison to CR; and Aim 3: To establish that ADMF is an effective diet therapy to maintain weight loss and sustain improvements in CHD risk indicators, and to compare changes in cognitive and behavioral components of eating between ADMF and CR subjects. A 52-week randomized, controlled, parallel-arm feeding trial will be implemented to test these objectives. The trial will be divided into 3 consecutive intervention periods: (1) 4-week baseline; (2) 24-week weight loss with food provided; and (3) 24-week weight maintenance with no food provided. Overweight and obese subjects (n = 90) will be randomized to 1 of 3 groups: (1) ADMF, 75% energy restriction on the "fast day" and ad libitum fed on the "feed day"; (2) CR, 25% restriction everyday; or 3) control, 100% energy intake everyday. During the weight maintenance phase, ADMF subjects will consume 25% of their energy needs on the "fast day" and 175% of their needs on the "feed day", while CR and control subjects will consume 100% of their needs everyday. Our findings will show that ADMF can be implemented as an alternative to CR to help overweight and obese individuals lose weight, maintain weight loss, and sustain reductions in CHD risk. This study will also generate insights into the specific behavioral changes that occur with ADMF that explain why ADMF is a successful diet strategy for weight maintenance.

ELIGIBILITY:
Inclusion criteria. Adult subjects meeting the following criteria will be eligible to participate:

* Age between 18 to 65 years old
* BMI between 25.0 and 39.9 kg/m2
* Previously sedentary (<60 minutes/week of light activity corresponding to 2.5 to 4.0 metabolic equivalents (METs) for the 3 months prior to the study)

Exclusion criteria. Subjects excluded from participating in the study include those who:

* Have a history cardiovascular disease (prior angina, myocardial infarction or stroke)
* Are diabetic (fasting blood glucose > 126 mg/dl)
* Have a history of psychiatric disorders and/or eating disorders
* Are taking anti-depressant or anti-anxiety medications
* Are taking drugs that affect study outcomes (weight loss, lipid-lowering, or blood pressure drugs)
* Are not weight stable for 3 months prior to the beginning of study (weight gain or loss > 4 kg)
* Are not able to keep a food diary or activity log for 7 consecutive days during screening
* Are perimenopausal or have an irregular menstrual cycle (menses that does not appear every 27-32 days)
* Are claustrophobic or have implanted electrical devices (cardiac pacemaker or a neurostimulator)
* Are pregnant, or trying to become pregnant
* Are smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krista Varady, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois, Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Lin S, Lima Oliveira M, Gabel K, Kalam F, Cienfuegos S, Ezpeleta M, Bhutani S, Varady KA. Does the weight loss efficacy of alternate day fasting differ according to sex and menopausal status? Nutr Metab Cardiovasc Dis. 2021 Feb 8;31(2):641-649. doi: 10.1016/j.numecd.2020.10.018. Epub 2020 Oct 31. PMID 33358713
- [Derived] Gabel K, Kroeger CM, Trepanowski JF, Hoddy KK, Cienfuegos S, Kalam F, Varady KA. Differential Effects of Alternate-Day Fasting Versus Daily Calorie Restriction on Insulin Resistance. Obesity (Silver Spring). 2019 Sep;27(9):1443-1450. doi: 10.1002/oby.22564. Epub 2019 Jul 22. PMID 31328895
- [Derived] Miranda ER, Fuller KNZ, Perkins RK, Kroeger CM, Trepanowski JF, Varady KA, Haus JM. Endogenous secretory RAGE increases with improvements in body composition and is associated with markers of adipocyte health. Nutr Metab Cardiovasc Dis. 2018 Nov;28(11):1155-1165. doi: 10.1016/j.numecd.2018.07.009. Epub 2018 Aug 2. PMID 30297199
- [Derived] Trepanowski JF, Kroeger CM, Barnosky A, Klempel M, Bhutani S, Hoddy KK, Rood J, Ravussin E, Varady KA. Effects of alternate-day fasting or daily calorie restriction on body composition, fat distribution, and circulating adipokines: Secondary analysis of a randomized controlled trial. Clin Nutr. 2018 Dec;37(6 Pt A):1871-1878. doi: 10.1016/j.clnu.2017.11.018. Epub 2017 Dec 5. PMID 29258678
- [Derived] Trepanowski JF, Kroeger CM, Barnosky A, Klempel MC, Bhutani S, Hoddy KK, Gabel K, Freels S, Rigdon J, Rood J, Ravussin E, Varady KA. Effect of Alternate-Day Fasting on Weight Loss, Weight Maintenance, and Cardioprotection Among Metabolically Healthy Obese Adults: A Randomized Clinical Trial. JAMA Intern Med. 2017 Jul 1;177(7):930-938. doi: 10.1001/jamainternmed.2017.0936. PMID 28459931

RESULTS

PARTICIPANT FLOW:
Groups:
- Alternate Day Fasting (ADF): Fast day diet: 25% energy intake, Feast day diet: Ad libitum energy intake (alternating days)
  Alternate day fasting
- Calorie Restriction (CR): 75% energy intake every day
  Calorie restriction
- Control: Usual diet
  Control diet
Period: Overall Study
Arm/Group | Alternate Day Fasting (ADF) | Calorie Restriction (CR) | Control
Started | 34 | 35 | 31
Completed | 21 | 25 | 23
Not Completed | 13 | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alternate Day Fasting (ADF) | Calorie Restriction (CR) | Control | Total
Number analyzed (Participants) | 34 | 35 | 31 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44 (10) | 43 (12) | 44 (11) | 44 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 27 | 86
  Male | 4 | 6 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 32 | 34 | 31 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 22 | 21 | 20 | 63
  White | 11 | 13 | 11 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: Change in body weight from baseline to month 12
Time Frame: Baseline to month 12
Measure: Mean (Standard Error); unit: Percent change at month 12
Arm/Group | Alternate Day Fasting (ADF) | Calorie Restriction (CR) | Control
Number analyzed (Participants) | 34 | 35 | 31
Percent change at month 12 | -4.6 (0.9) | -4.5 (0.9) | 0.3 (0.6)

2. Secondary Outcome: Change in HDL Cholesterol
Description: Change in HDL cholesterol from baseline to month 12
Time Frame: 12 month interval
Measure: Mean (Standard Error); unit: Percent change from baseline to month 12
Arm/Group | Alternate Day Fasting (ADF) | Calorie Restriction (CR) | Control
Number analyzed (Participants) | 34 | 35 | 31
Percent change from baseline to month 12 | 4.6 (3.1) | -0.5 (3.1) | -3.4 (3.9)

3. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure from baseline to month 12
Time Frame: 12 month interval
Measure: Mean (Standard Error); unit: Percent change from baseline to month 12
Arm/Group | Alternate Day Fasting (ADF) | Calorie Restriction (CR) | Control
Number analyzed (Participants) | 34 | 35 | 31
Percent change from baseline to month 12 | -3.5 (2.3) | -2.9 (2.0) | -2.6 (4.0)

4. Secondary Outcome: Change in Fasting Glucose
Description: Change in fasting glucose from baseline to month 12
Time Frame: 12 month interval
Measure: Mean (Standard Error); unit: Percent change from baseline to month 12
Arm/Group | Alternate Day Fasting (ADF) | Calorie Restriction (CR) | Control
Number analyzed (Participants) | 34 | 35 | 31
Percent change from baseline to month 12 | 4.0 (2.0) | -1.9 (3.3) | 10.7 (3.4)

5. Secondary Outcome: Change in Fasting Insulin
Description: Change in fasting insulin from baseline to month 12
Time Frame: 12 month interval
Measure: Mean (Standard Error); unit: Percent change from baseline to month 12
Arm/Group | Alternate Day Fasting (ADF) | Calorie Restriction (CR) | Control
Number analyzed (Participants) | 34 | 35 | 31
Percent change from baseline to month 12 | -35 (11) | -28 (9) | -2.5 (13)

6. Secondary Outcome: Change in Insulin Resistance Measured by HOMA-IR
Description: Change in insulin resistance measured by HOMA-IR from baseline to month 12
Time Frame: 12 month interval
Measure: Mean (Standard Error); unit: Percent change from baseline to month 12
Arm/Group | Alternate Day Fasting (ADF) | Calorie Restriction (CR) | Control
Number analyzed (Participants) | 34 | 35 | 31
Percent change from baseline to month 12 | -36 (13) | -34 (12) | 12 (16)

7. Secondary Outcome: Change in Plasma C-reactive Protein Concentrations
Description: Change in plasma C-reactive protein concentrations from baseline to month 12
Time Frame: 12 month interval
Measure: Mean (Standard Error); unit: Percent change from baseline to month 12
Arm/Group | Alternate Day Fasting (ADF) | Calorie Restriction (CR) | Control
Number analyzed (Participants) | 34 | 35 | 31
Percent change from baseline to month 12 | -13.9 (11.7) | -6.2 (8.1) | 5.4 (16.8)

8. Secondary Outcome: Change in Plasma Homocysteine Concentrations
Description: Change in plasma Homocysteine concentrations from baseline to month 12
Time Frame: 12 month interval
Measure: Mean (Standard Error); unit: Percent change from baseline to month 12
Arm/Group | Alternate Day Fasting (ADF) | Calorie Restriction (CR) | Control
Number analyzed (Participants) | 34 | 35 | 31
Percent change from baseline to month 12 | 0.2 (4.3) | -1.2 (3.2) | -2.6 (3.3)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Alternate Day Fasting (ADF) | Calorie Restriction (CR) | Control
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35 | 0/31
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35 | 0/31

LIMITATIONS AND CAVEATS:
1. The duration of the maintenance phase was short (6 months).
2. The dropout rate was higher than anticipated.
3. We enrolled predominantly metabolically healthy obese individuals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No